CLINICAL TRIAL: NCT04046250
Title: Phase 2a, Multi-center, Placebo-controlled, Randomized, Partially Blinded, Study Infused TK112690 or or Placebo Administered Along With Methotrexate Weekly for Four Consecutive Weeks to Patients With Recurrent or Residual SCCHN
Brief Title: Phase 2a Study to Evaluate Suppression of Methotrexate-induced Mucositis by TK112690
Acronym: TK112690
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tosk, Inc. (Industry)
Collaborators: Crystal Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLP-2690-0003
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Results first posted 2021-06-03 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Mucositis
Keywords: Mucositis; Methotrexate; Uridine Phosphorylase Inhibitor; Head and Neck Cancer
MeSH Terms: conditions — Mucositis; Head and Neck Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: A total of 22 patients will be enrolled into one of 2 different: TK112690 treated or placebo treated.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study will be partially blinded. The patient and investigator will be blinded as to whether TK112690 or placebo is administered. The clinical research organization, sponsor, and site pharmacist will know whether the patient was administered active drug or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- TK112690 (Experimental): TK112690 treatment
  Interventions: Drug: TK-112690
- Placebo (Placebo Comparator): TK112690 formulation
  Interventions: Drug: Placebo TK-112690

INTERVENTIONS:
Drug: TK-112690 — TK112690 treatment pre-methotrexate treatment
  Other Names: Treatment
  Arms: TK112690
Drug: Placebo TK-112690 — Placebo
  Arms: Placebo

SUMMARY:
Patients will receive methotrexate at a dose of 45 mg/m2 administered weekly for 4 consecutive weeks as an iv infusion along with a nutritional supplement administered two hours before the methotrexate. One hour before the methotrexate treatment the patients will be administered the first infusion of the day of either TK112690 or placebo depending on randomization. Five hours after the methotrexate treatment the patients will be administered the second treatment of either TK112690 or placebo depending on randomization. The TK112690 dose will be 45 mg/kg.

DETAILED DESCRIPTION:
Patients will receive methotrexate at a dose of 45 mg/m2 administered weekly for 4 consecutive weeks as an iv infusion along with a nutritional supplement administered two hours before the methotrexate. One hour before the methotrexate treatment the patients will be administered the first infusion of the day of either TK112690 or placebo depending on randomization infusion. Five hours after the methotrexate treatment the patients will be administered the second treatment of either TK112690 or placebo depending on randomization. The TK112690 dose will be 45 mg/kg.

* A total of 22 patients will be enrolled into one of 2 different dose groups: TK-112690 treated or placebo treated.
* Screening must be within 15 days of subject enrollment.
* Patients will remain for observation at the clinical site for a minimum of 25 hours post initial TK112690 or placebo dose.
* Study follow-up will occur on Week 6, two weeks after the last dosing of methotrexate.
* Blinding: The study will be partially blinded. The patient and investigator will be blinded as to whether TK112690 or placebo is administered. The CRO, sponsor, and site pharmacist will know whether the patient was administered active drug or placebo.

ELIGIBILITY:
Inclusion Criteria

* Male and female subjects over 18 years old with a histologically or cytological confirmed diagnosis of locally residual, recurrent or metastatic SCCHN.
* Subject must have failed at least one courses of non-MTX chemotherapy, or one course of non-MTX chemotherapy and chemo radiation for treating their SCCHN.
* No prior systemic treatments for cancer (chemotherapy and/or radiotherapy) 4 weeks prior to screening.
* No other concurrent, active, invasive malignancies.
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Must have a life expectancy of at least 6 months.
* History of brain metastases allowed if disease has stabilized or improved after radiation and/or craniotomy.
* No active angina or uncontrolled arrhythmia.
* No detectable infection including hepatitis B/C and HIV.
* Not pregnant or nursing. Women of childbearing potential must have a negative urine pregnancy test at screening and on the day before dosing and must use medically acceptable methods of birth control. Acceptable methods of birth control include oral or transdermal contraceptives, condoms, spermicidal foam, IUD, progestin implant or injection, abstinence, vaginal ring, or sterilization of partner. The reason for non-childbearing potential, such as bilateral tubal ligation, bilateral oophorectomy, hysterectomy, or post-menopausal for ≥ 1 year, must be specified in the patient's medical history file and CRF.
* Must have adequate organ and immune function as indicated by the following laboratory values:

Parameter Laboratory Values Serum creatinine ≤1.5 x ULN Est. creatinine clearance ≥45 mL/min Total bilirubin ≤2.0 mg/dL (≤34.2 μmol/L) AST & ALT ≤3 x ULN Absolute granulocytes ≥1.5 x 109 cells/L Platelets ≥100,000/µL

● Be able to read and understand, and provide a signature or thumb impression on the Informed Consent Form (ICF) before entering the study.

Exclusion Criteria:

* Subject has not failed at least one courses of non-MTX chemotherapy or one course of non-MTX chemotherapy and chemo radiation for treating their SCCHN.
* Uncontrolled active infection.
* Current mucositis (>Grade 1).
* Pregnant or nursing mother.
* Prior history of a cerebrovascular accident or hemorrhage.
* Congestive heart failure, as defined by New York Heart Association class III or IV.
* Uncontrolled hypertension.
* Active psychiatric/mental illness making informed consent or useful clinical follow-up unlikely.
* Subjects who have previously been enrolled into this study and subsequently withdrew.
* Subject receiving other investigational agent(s).
* Any systemic immunosuppressive medication/therapy (eg, other chemotherapy, steroids).
* Any significant systemic illness, unstable or severe medical condition(s) that could put the subject at risk during the study, interfere with outcome measures, or affect compliance with the protocol procedures such as intercurrent infection and/or autoimmune disease, ie, any condition that compromises the immune system.
* Known or suspected intolerance or hypersensitivity to the study materials (TK-112690 and/or excipients or closely related compounds).
* Subjects, who have received, or plan to receive, radiation or chemotherapy within 4 weeks of screening.
* Subjects that have a history of poor compliance in clinical research studies.
* Subjects that have participated in any other investigative clinical trial in the past 4 weeks.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emile Youssef, MD, PhD, Study Director — Tosk, Inc.
Locations (3):
- India (3):
  - Bangalore Cancer, Bangalore, Karnataka
  - Karnatak Cancer Therapy and Research Institute, Navanagar, Karnataka
  - Netaji Subhash Chandra Bose Cancer Hospital, Kolkata, West Bengal

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TK112690 | Placebo
Started | 11 | 11
Completed | 8 (Four Methotrexate + TK-112690 Treatments) | 7 (Four Methotrexate + TK-12260 Placebo Treatments)
Not Completed | 3 | 4
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TK112690 | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11) | 49 (13) | 52 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mucositis
Description: Mucositis Evaluation Using Established Scoring Systems: NCI/CTCAE at 4 WKs (Primary) and WHO at 4 WKs (Primary).
  NCI/CTCAE=National Cancer Institute/Common Terminology Criteria for Adverse Events and WHO=World Health Organization
  NCI Grades- 0= No mucositis, 1=Mild mucositis (Painless ulcers, erythema, or mild soreness in the absence of lesions), 2=Moderate mucositis (Painful erythema, edema, or ulcers but eating or swallowing possible), 3= Severe mucositis (Painful erythema, edema, or ulcers requiring IV hydration), 4=Life threatening, 5=Death WHO Grades- 0=No mucositis, 1= Mild (Oral soreness, erythema), 2=Moderate (Oral erythema, ulcers, solid diet tolerated), 3=Severe (Oral ulcers, liquid diet only), 4=Life-threatening (Oral alimentation impossible).
  For both the scales above, a higher score implies greater mucositis.
  Scale specific mean values for patients in each group (placebo or treated) are calculated and compared by Student's t-test.
Time Frame: up to 4 Weeks
Population: Patients with SCCHN who have failed at least one prior treatment of chemotherapy and/or radiation
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TK112690 | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale
  NCI/CTCAE at 4 WKs: number analyzed (Participants) | 8 | 7
  NCI/CTCAE at 4 WKs | 0.37 (0.19) | 2.84 (0.29)
  WHO at 4 WKs: number analyzed (Participants) | 8 | 7
  WHO at 4 WKs | 0.34 (0.17) | 2.87 (0.31)

2. Secondary Outcome: Incidence Adverse Events That Are Related to Treatment
Description: Tolerance
Time Frame: Measured Weekly Over 4 Weeks of Study
Measure: Count of Participants; unit: Participants
Arm/Group | TK112690 | Placebo
Number analyzed (Participants) | 11 | 11
Participants
  SAEs | 0 | 2
  Deaths | 0 | 1
  TEAE GI and Related | 1 | 11

ADVERSE EVENTS:
Time Frame: 6 Weeks
Arm/Group | TK112690 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 2/11
Other Adverse Events (participants affected / at risk) | 1/11 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TK112690 (N=11) | Placebo (N=11)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TK112690 (N=11) | Placebo (N=11)
GI Disorders (Gastrointestinal disorders) | 1 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each of the three clinical sites has a PI. Each PI is bound by a CDA covering the clinical data.

Tosk intends to prepare a manuscript reporting results from this trial combined with the results from the Phase 1b clinical trial. All the PIs will have a chance to review and approve the findings reported in the manuscript. Tosk expects to submit the manuscript for publication in early 2022.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/50/NCT04046250/Prot_SAP_000.pdf